CLINICAL TRIAL: NCT04830319
Title: Therapeutic Effect of the Pilates Method in People With HAM/TSP: a Randomized Crossover Study
Brief Title: Pilates Method in People With HAM/TSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedreira, Érika, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HTLVIDA
Record Dates: First submitted 2018-05-23; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: HAM/TSP; HTLV-1 Secondary Myelopathy; Balance; Gait Balance; Functional Mobility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test-control group (TCG) (Experimental): The test-control group (TCG) will initiate the protocol with exercises of the Pilates method, which includes exercises in soil, that associate the correct respiratory movement with muscular strengthening and control, stretching from the eccentric movement, selective upper and lower trunk movements. There will be used accessories described by the method for their realization. Participants will perform the first week of awareness and body alignment exercises for 10 minutes, 10 minute breath perception, 10 minute proximal muscle accuracy and control, and 10 minute stretches; from the second week will be included selective trunk movements, with muscle strengthening of lower limbs. Rest intervals will be performed between exercises.After 20 sessions, the patients will be reassessed and will remain for a period of one month without any intervention, and at the end of this period will be reevaluated again. The TCG group will then conduct 20 task-oriented training sessions
  Interventions: Other: Pilates Method; Other: task-oriented training protocol
- Control-test group (CTG) (Active Comparator): The control-test group (CTG) will initiate the task-oriented training protocol. The task-oriented training protocol will include functional exercise drills, such as sit-up and workout, obstacle course workout, speed-and-direction workout, balance workout, work-up and downhill workout, each tasks performed for eight minutes, with two minutes of rest between them. The difficulty in carrying out the tasks will be progressively adjusted. At all times, individuals will be instructed to contract the pelvic floor musculature. After 20 sessions, the patients will be reassessed and will remain for a period of one month without any intervention, and at the end of this period will be reevaluated again. Next, the CTG group will perform 20 sessions of Pilates exercises.
  Interventions: Other: Pilates Method; Other: task-oriented training protocol

INTERVENTIONS:
Other: Pilates Method — includes exercises in soil, that associate the correct respiratory movement with muscular strengthening and control, stretching from the eccentric movement, selective upper and lower trunk movements. There will be used accessories described by the method for their realization. Participants will perform the first week of awareness and body alignment exercises for 10 minutes, 10 minute breath perception, 10 minute proximal muscle accuracy and control, and 10 minute stretches; from the second week will be included selective trunk movements, with muscle strengthening of lower limbs. Rest intervals will be performed between exercises.
Other: task-oriented training protocol — The control-test group (CTG) will initiate the task-oriented training protocol. The task-oriented training protocol will include functional exercise drills, such as sit-up and workout, obstacle course workout, speed-and-direction workout, balance workout, work-up and downhill workout, each tasks performed for eight minutes, with two minutes of rest between them. The difficulty in carrying out the tasks will be progressively adjusted. At all times, individuals will be instructed to contract the pelvic floor musculature. After 20 sessions, the patients will be reassessed and will remain for a period of one month without any intervention, and at the end of this period will be reevaluated again. Next, the CTG group will perform 20 sessions of Pilates exercises.

SUMMARY:
Individuals with HTLV-1 secondary myelopathy (HAM/TSP) may have motor and sensory alterations, which may result in reduced functional performance and consequent risk of falls. The aim of the study is to verify the therapeutic effect of a Pilates exercise program on functional performance and risk of falls, when compared to task-oriented training, of people with HAM / TSP. This is a randomized, crossover clinical trial performed with individuals with HAM / TSP who are attended at a referral center who is able to perform gait whether or not to use a walking aid. Amputees, with psychiatric disorders, rheumatic or orthopedic diseases and other associated neurological disorders, which could influence the balance and functional mobility, as well as pregnant women, were excluded. Participants will be submitted to the initial evaluation of functional mobility, balance, gait balance, fatigue, gait endurance, sphincter changes and questioned about the occurrence of falls in the last three months and will answer a semi-structured questionnaire about their conjugality. They will be allocated randomly to two groups. One will perform the Pilates Method protocol and the other task-oriented training. The first group, called test-control group (GTC), will initiate the protocol with exercises of the Pilates method; the control-test group (GCT) will initiate the task-oriented training protocol. A p <0.05 will be considered a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* individuals with probable and/or defined diagnosis of HAM / TSP, according to WHO criteria, of both sexes, aged 18 to 64 years.

Exclusion Criteria:

* individuals with lower limb amputation, pregnancy, psychiatric disorders, rheumatic or orthopedic diseases, other associated neurological disorders, and those who have difficulty understanding the assessment instruments.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Balance | 15 minutes
  Berg's Balance Scale (BBS)
Functional Mobility | 3 minutes
  Timed up and Go (TUG)
Gait Balance | 10 minutes
  Dynamic Gait Index (DGI)
Balance | 20 minutes
  Balance Evaluation Systems Test of dynamic balance (mini-BESTest)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Católica do Salvador, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No